CLINICAL TRIAL: NCT04152291
Title: The Effect of Ethyl Eicosapentaenoic Acid on Circulating Low-density Lipoproteins and Plasma Lipid Metabolism in Healthy Volunteers
Brief Title: The Effect of E-EPA on Circulating LDL and Plasma Lipid Metabolism
Acronym: EPA&LDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wihuri Research Institute (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Katariina Öörni, Group leader, Professor, Ph. D, Wihuri Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E-EPA
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Atherosclerosis; Low-density Lipoproteins Aggregation Susceptibility; Low-density Lipoprotein Lipid Composition; Cardiovascular Diseases
Keywords: Atherosclerosis; E-EPA; LDL aggregation susceptibility; Lipidomics; Proteoglycan binding; Icosapent ethyl; Fatty acid; Metabolism; Omega-3
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Intervention Model Description: Baseline measurements are compared to different time points during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-EPA-diet group (Experimental): All the study participants will receive the same treatment. 3.9g of E-EPA in capsules, which also include 75µg of D3-vitamin, daily for 28 days.
  Interventions: Dietary Supplement: Ethyl-Eicosapentaenoic Acid (E-EPA)

INTERVENTIONS:
Dietary Supplement: Ethyl-Eicosapentaenoic Acid (E-EPA) — 3,9 grams of E-EPA (Icosapent ethyl) is added to participants' normal diet.
  Other Names: E-EPA; Icosapent ethyl

SUMMARY:
40-70 healthy volunteers of ages 18 to 65 participate in a E-EPA-diet where 3,9 grams of E-EPA is added to their normal diet and lifestyles for a month. Blood samples will be collected before the study and at weeks 1 and 4 and also, two weeks after finishing the diet. Main study focuses are LDL aggregation susceptibility, lipid composition and proteoglycan binding affinity. In addition, important plasma lipid metabolism enzymes and lipid mediated resolvins are measured as well as several baseline characteristics.

DETAILED DESCRIPTION:
Four grams of daily E-EPA was found to significantly decrease atherosclerotic cardiovascular diseases in the REDUCE-IT study. In the upcoming study the effect of E-EPA to low-density lipoprotein (LDL) aggregation susceptibility is measured using dynamic light scattering technique to continuously measure particles size while inducing aggregation. LDL Lipid composition is analyzed using electrospray mass spectrometer optimized for lipid measurements. Previously is reported that the aggregation susceptibility is affected by the lipid composition which is modifiable (Ruuth et. al. Eur.H.Journal 2018). Common disease factors such as total cholesterol, LDL, HDL, triglycerides, ApoB-100, ApoA-I, Lp(a) and different modified LDL levels are measured. Also, activities of lipid metabolism enzymes like PON-1, LCAT, CETP, PLTP and lipid mediated resolvins are looked into. Objective is to identify changes and possible pathways that are altered by the increase of E-EPA and to use the data to possibly explain the health benefits of EPA.

Update at study conclusion 17.6.2025. Covid-19 halted our study progression leading to a partial cohort (final n=38). Covid-19 restrictions also prevented us from measuring plasma lipid metabolism enzymes and lipid mediated resolvins. As a results we expanded the lipoprotein lipidomics analysis to consist all three lipoprotein fractions (VLDL, LDL, and HDL) using LC/MS. Finally a clinical cardiovascular risk score assessment was also performed (CERT2/Hertta-test).

ELIGIBILITY:
Inclusion Criteria:

* Healthy normolipidemic

Exclusion Criteria:

* Prescription of blood thinner medicine
* Circulating Low-density lipoprotein > 5mmol/l, Triglycerides >3mmol/l
* Chronic use of pain medication
* Fish allergy
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katariina Öörni, Professor, Ph.D, Principal Investigator — Wihuri Research Institute
Locations (1):
- Wihuri Research Institute, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in compliance with EU's General Data Protection Regulation (GDPR)

REFERENCES:
- [Background] Ruuth M, Nguyen SD, Vihervaara T, Hilvo M, Laajala TD, Kondadi PK, Gistera A, Lahteenmaki H, Kittila T, Huusko J, Uusitupa M, Schwab U, Savolainen MJ, Sinisalo J, Lokki ML, Nieminen MS, Jula A, Perola M, Yla-Herttula S, Rudel L, Oorni A, Baumann M, Baruch A, Laaksonen R, Ketelhuth DFJ, Aittokallio T, Jauhiainen M, Kakela R, Boren J, Williams KJ, Kovanen PT, Oorni K. Susceptibility of low-density lipoprotein particles to aggregate depends on particle lipidome, is modifiable, and associates with future cardiovascular deaths. Eur Heart J. 2018 Jul 14;39(27):2562-2573. doi: 10.1093/eurheartj/ehy319. PMID 29982602
- [Background] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Cardiovascular Risk Reduction with Icosapent Ethyl for Hypertriglyceridemia. N Engl J Med. 2019 Jan 3;380(1):11-22. doi: 10.1056/NEJMoa1812792. Epub 2018 Nov 10. PMID 30415628
- [Result] Preprint/ Lauri Äikäs, Petri T. Kovanen, Martina Lorey, Reijo Laaksonen, Minna Holopainen, Hanna Ruhanen, Reijo Käkelä, Matti Jauhiainen, Martin Hermansson, Katariina Öörni. Remodelling of plasma lipoproteins by icosapent ethyl -supplementation and its impact on cardiovascular disease risk markers in normolipidemic individuals. MedRxiv 2024.11.27.24318042; doi: https://doi.org/10.1101/2024.11.27.24318042
- See also: Preprint of the research article from the study — https://www.medrxiv.org/content/10.1101/2024.11.27.24318042v1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in autumn/winter of 2019/2020 via in-house emailing lists. Participant suitability was assessed prior to the beginning of the supplementation. Healthy normolipidemic individuals aged 18-65 were enrolled.
Groups:
- IPE-supplementation Group: All the study participants will receive the same treatment. 3.9g of IPE (Ethyl-EPA) in capsules, which also include 75µg of D3-vitamin, daily for 28 days.
Period: Overall Study
Arm/Group | IPE-supplementation Group
Started | 68
Completed | 38
Not Completed | 30
Not completed — Covid-19 restrictions | 27
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Final number included in the analyses
Arm/Group | IPE-supplementation Group
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 38
LDL-cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.7 (0.4)
Blood triglycerides [Mean (Standard Deviation); unit: mmol/L] | 0.9 (0.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 23.5 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: LDL Aggregation Susceptibility
Description: LDL aggregation susceptibility was induced in vitro by sphingomyelinase and measured using dynamic light scattering. Time-size curves were generated, and the inflection point (EC50)-the midpoint of the most rapid aggregation-was determined by nonlinear regression with a modified Hill equation. A longer time to reach EC50 indicates lower aggregation susceptibility, and thus a lower risk of future cardiovascular events.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- IPE-supplementation Group: All the study participants will receive the same treatment. 3.9g of IPE (Ethyl-EPA) in capsules, which include 75µg of D3-vitamin, daily for 28 days.
Arm/Group | IPE-supplementation Group
Number analyzed (Participants) | 38
Minutes
  Baseline | 111.3 (17.3)
  After 28-day of IPE-supplementation | 113.1 (25.8)

2. Primary Outcome: Total Blood Triglycerides
Description: Percentage change in blood triglycerides after IPE-supplementation (day 28) compared to the baseline (day 0). Percentage change was calculated as follows: [(day 28 - day 0) / day 0] x 100.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage of baseline triglycerides
Arm/Group | IPE-supplementation Group
Number analyzed (Participants) | 38
percentage of baseline triglycerides | -14 (28)

3. Primary Outcome: EPA Incorporation Into LDL
Description: Total concentration of eicosapentaenoic acid in LDL lipoprotein fraction at baseline (day 0), and after IPE-supplementation (day 28).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IPE-supplementation Group
Number analyzed (Participants) | 38
mmol/L
  Baseline | 0.075 (0.094)
  After 28-day of IPE-supplementation | 0.274 (0.118)

4. Other Pre Specified Outcome: Lipoprotein Retention
Description: The binding of lipoproteins to aortic proteoglycans, measured ex vivo. At the end of the assay lipoprotein-associated bound cholesterol is measured in each well and compared to control wells to determine the binding probability of LDL particles to aortic proteoglycans.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Bound cholesterol nmol/well
Arm/Group | IPE-supplementation Group
Number analyzed (Participants) | 38
Bound cholesterol nmol/well
  Baseline | 4.995 (0.041)
  After 28-day of IPE-supplementation | 4.428 (0.039)

5. Other Pre Specified Outcome: Coronary Event Risk Test 2
Description: A clinical risk rest used to assess 10-year Coronary event risk. Based on plasma ceramides and phospholipids. Lower risk score indicates smaller future risk of coronary events. The four risk categories are: 0-3 (Low risk), 4-6 (Moderate risk), 7-8 (High risk), and 9-12 (Very high risk).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IPE-supplementation Group
Number analyzed (Participants) | 38
Scores on a scale
  Baseline | 3.4 (2.6)
  After 28-day of IPE-supplementation | 2.5 (1.8)

ADVERSE EVENTS:
Time Frame: From enrollment until the end of the washout period (35 days)
Arm/Group | IPE-supplementation Group
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

LIMITATIONS AND CAVEATS:
Covid-19 halted the study. This study's small sample size and focus on normolipidemic, Finnish, white Caucasian volunteers may limit its generalization to broader populations. The IPE preparation contained vitamin D3, which can influence plasma lipoprotein profiles, although it's kinetics differ from most measured parameters. The study's short duration also prevents assessment of IPE's long-term effects on lipoprotein profiles and cardiovascular outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04152291/Prot_SAP_ICF_000.pdf